CLINICAL TRIAL: NCT05178511
Title: a Prospective, Open Phase ii Clinical Study in Patients With alK-positive Non-small Cell Lung Cancer Treated With Ensatinib After Second-generation ALK-TKI Resistance
Brief Title: Ensatinib Treat Second-generation ALK-TKI Resistance After Second-generation ALK-TKI Resistance
Acronym: ERSGATR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, MD, head of department, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV001
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: The Diagnosis Was ALK Positive NSCLC; Second Generation ALK-TKI is Resistant; Efficacy of Ensatinib in This Subset of Patients
Keywords: ensartinib
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hydrochloric acid ensartinib (Experimental): Ensatinib 225mg daily, QD, until progression or intolerance
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Ensaritinib was taken orally once 225mg, on an empty stomach or with food, until the patient developed disease progression, developed unacceptable toxicity, the investigator or subject decided to drop out, lost follow-up, initiated other antitumor therapy, or died
  Other Names: X-396

SUMMARY:
After the use of second-generation ALK-TKI drug resistance, about 50% of tissue biopsies showed mutations in the ALK kinase domain, and appropriate ALK-TKI could be selected according to different mutation sites .Phase I/II clinical trials in the US of ensatinib showed ORR of 25% (4/16) in patients previously treated with crizotinib and second-generation ALK-TKI (N=16) .In the phase II registered clinical study in China, biomarker analysis also showed that the ORR of ensatinib against drug resistance site G1202R was 33% (2/6).The ORR of I1171 and F1174 were 50% (2/4) and 71% (5/7), respectively, suggesting that ensatinib may still be effective in patients with drug resistance to other second-generation ALK inhibitors . Investigators designed this study to evaluate the clinical efficacy of ensatinib after second-generation ALK-TKI resistance.The study was a single-arm, multi-center Phase II clinical study, using ORR of patients with measurable lesions as the primary endpoint, and using Simon two-stage design to estimate the required sample size.At a 5% level of significance and 85% confidence, a minimum of 40 evaluable subjects were required for both phases.In the first stage, 20 patients were enrolled. If 2 patients had objective response, an additional 20 patients were enrolled in the second stage. If more than 5 patients /40 patients had objective response, the therapeutic drugs were considered effective.Eligible patients will take 225mg of ensaritinib orally once daily, on an empty stomach or with food, until the patient develops disease progression, develops unacceptable toxicity, the investigator or subject decides to drop out, loses follow-up, starts another antitumor therapy, or dies.The primary end points were objective response rate (ORR) to disease progression, occurrence of unacceptable toxicity, investigator or subject decision to drop out, loss of follow-up, initiation of other antitumor therapy, or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) confirmed histologically or cytologically ;
* Patients confirmed as ALK positive (FISH or Ventana IHC or RT-PCR, NGS) in previous written reports.Disease progression after continuing treatment with prior second-generation ALK-TKI resistance (allowing crizotinib resistance) (as per RECIST 1.1);
* Maximum one chemotherapy is allowed;The interval between the last administration of second-generation ALK-TKI and the trial enrollment should be at least 7 days;
* Gender: both male and female;Age: ≥18 years old;
* physical status score was 0-2;
* survival ≥3 months;
* certain organ system functions (no blood transfusion or use of constituent blood within 14 days before test)；
* Asymptomatic CNS metastases that do not require treatment with steroids or anticonvulsants;If there is CNS metastasis, radiotherapy can be performed first, and no progress can be made after ≥28 days.Meningeal disease was not included in the group;
* Patients must have measurable lesions according to RECIST1.1 criteria;
* Willing and able to follow the trial and follow-up procedures;
* Able to understand the nature of the experiment and sign written informed consent voluntarily.

Exclusion Criteria:

* Patients who had previously only used crizotinib or loratinib；
* Currently receiving other systemic anti-tumor treatments；
* history of malignancy other than lung cancer in the past 3 years (excluding cured basal cell tumor of the skin, early gastrointestinal [GI] tumor resected under endoscope, carcinoma in situ of the cervix)；
* Patients who participated in clinical trials of other investigational drugs within weeks prior to initial ensatinib administration；
* Major surgery or immunotherapy within 4 weeks prior to initial; dosing;Radiation therapy was received within 2 weeks prior to initial dosing；
* In the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results;
* Other conditions considered unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 0 up to 8 weeks

SECONDARY OUTCOMES:
Progression free survival | 0 up to12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code